CLINICAL TRIAL: NCT04487028
Title: Dysphagia in Thoracic Surgical Patients: Incidence, Risk-factors, and Health Related Outcomes
Brief Title: Dysphagia in Thoracic Surgical Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202000724-A
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Thoracic Diseases
Keywords: Dysphagia; Extubation; Vocal Fold Mobility Impairment; Peak Cough Flow (PCF)
MeSH Terms: conditions — Thoracic Diseases; Deglutition Disorders | interventions — Fees and Charges

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic Surgical Patients: Participants will undergo a Fiberoptic Endoscopic Evaluation of Swallowing (FEES)
  Interventions: Procedure: Fiberoptic Endoscopic Evaluation of Swallowing

INTERVENTIONS:
Procedure: Fiberoptic Endoscopic Evaluation of Swallowing — This procedure involves inserting a flexible laryngoscope that contains a light source and video camera on the end through the open passage of the nose towards the back of the throat in order to visualize the swallowing mechanism.
  Other Names: FEES

SUMMARY:
The proposed study seeks to determine the incidence of dysphagia and vocal fold mobility impairment (VFMI) in individuals undergoing throacic surgical procedures. It also seeks to determine the impact of postoperative swallowing impairment on health-related outcomes.

DETAILED DESCRIPTION:
Swallowing impairment and VFMI are common, yet often overlooked, complications of thoracic surgical procedures. The true incidence of both dysphagia and VFMI in this patient population is unclear due to a lack of rigorous study using instrumental assessment techniques and validated outcomes in all patents undergoing thoracic surgery. The study is therefore aimed to determine the incidence of dysphagia and VFMI in this patient population and to characterize impairment profiles related to swallowing safety and efficiency. In addition, the study is also aimed to assess the relative impact of VFMI and dysphagia on health-related outcomes such as length of hospital stay, pneumonia, sepsis, reintubation, and discharge status

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 - 90 years old
* undergoing planned or emergent thoracic surgery via clamshell and/or extended thoracotomy
* confirmed negative COVID-19 test
* willing to participate in postoperative swallowing evaluation testing.

Exclusion Criteria:

* individuals under the age of 18.
* pregnant
* or those testing positive for COVID-19
* Additionally, the inability to demonstrate appropriate alertness and cognitive status following the procedure will exclude a participant from participating in this study to ensure protection of vulnerable individuals.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 240 individuals undergoing thoracic surgery will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | Baseline
  This scale is a validated measure used by trained blinded clinicians to assign ratings of safety to swallowing bolus trials. The development and use of an 8-point, equal-appearing interval scale (8 being best; 1 being worst) to describe penetration and aspiration events are described. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled.

SECONDARY OUTCOMES:
Yale Residue Severity Rating Scale | Baseline
  This scale is a validated measure used by trained blinded clinicians to assign ratings of efficiency to swallowing bolus trials. The Yale Pharyngeal Residue Severity Rating Scale was developed, standardized, and validated to provide reliable, anatomically defined, and image-based assessment of post-swallow pharyngeal residue severity as observed during fiberoptic endoscopic evaluation of swallowing (FEES). It is a five-point ordinal rating scale based on residue location (vallecula and pyriform sinus) and amount (none, trace, mild, moderate, and severe).

OTHER OUTCOMES:
Vocal Fold Mobility Impairment | Baseline
  During a Fiberoptic Endoscopic Evaluation of Swallowing (FEES), the vocal folds will be visualized using a small camera passed through the open nasal passage. The patient will be asked to make a series of vocal tasks so that we can visualize their movement, any immobility will be notated.

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Plowman, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Cardiovascular Clinic at UF Health UF, Gainesville, Florida
  - Thoracic and Cardiovasscular Surgery at UF Health, Gainesville, Florida
  - UF Health at the University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No